CLINICAL TRIAL: NCT01447537
Title: Mechanisms Involved in the Benefits of an Exercise Programme in Patients With Cirrhosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Principal Investigator, German Soriano, Dr. German Soriano Pastor Principal Investigator, Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IIBSP-PEF-2010-50
Record Dates: First submitted 2011-09-28; First posted 2011-10-06 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-12

CONDITIONS: Cirrhosis
Keywords: Cirrhosis; Exercise; Relaxation; Muscle mass; Effort tolerance
MeSH Terms: conditions — Fibrosis; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise, relaxation (Active Comparator): Active comparator: Exercise + relaxation Patients will perform exercise + relaxation for 3 months
  Interventions: Other: Exercise + relaxation
- Relaxation (Other): Relaxation without exercise Patients will receive only relaxation for 3 months
  Interventions: Other: Relaxation

INTERVENTIONS:
Other: Exercise + relaxation — Exercise + relaxation
  Arms: Exercise, relaxation
Other: Relaxation — Relaxation without exercise Patients will receive only relaxation for 3 months
  Arms: Relaxation

SUMMARY:
The investigators conducted a pilot study including 17 patients with liver cirrhosis showing that a moderate exercise programme during three months increased thigh circumference,exercise tolerance and quality of life without adverse effects. The present study aim to more accurately evaluate the effect of exercise on muscle mass, effort tolerance and inflammatory response in patients with cirrhosis. This study will include 30 patients with compensated liver cirrhosis that will be randomized into two groups: exercise group and control group. Evaluation of muscle mass, effort tolerance, inflammatory response and quality of life will be made at the beginning and at the end of the study.

DETAILED DESCRIPTION:
Exercise group: will do a physiotherapist supervised exercise programme 1 hour three times per week during three months and relaxation after exercise. Control group: only relaxation 1 hour three times per week during three months.

Assessment: clinical and laboratory examinations performed at baseline and at the end of the study. The investigators will analyze the changes in muscle mass by anthropometric measurements and advanced techniques (CT scan, densitometry), effort tolerance (stress test), quality of life (sF-36), glutamine synthetase activity in blood, oxidative damage and inflammatory response. The investigators will analyze the survival and complications of cirrhosis during the study and follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Compensated liver cirrhosis

Exclusion Criteria:

* hepatocellular carcinoma
* active alcoholism (less than 1 year)
* decompensated cirrhosis
* variceal bleeding less than 3 months.
* contraindication for exercise

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-09; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Increase in muscle mass | Basal and three months
Change in Effort tolerance | Basal and three months

CONTACTS AND LOCATIONS:
Overall Officials: German Soriano MD PhD, Principal Investigator — Department of Gastroenterology, Hospital de la Santa Creu i Sant Pau
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona, Spain

REFERENCES:
- [Derived] Roman E, Garcia-Galceran C, Torrades T, Herrera S, Marin A, Donate M, Alvarado-Tapias E, Malouf J, Nacher L, Serra-Grima R, Guarner C, Cordoba J, Soriano G. Effects of an Exercise Programme on Functional Capacity, Body Composition and Risk of Falls in Patients with Cirrhosis: A Randomized Clinical Trial. PLoS One. 2016 Mar 24;11(3):e0151652. doi: 10.1371/journal.pone.0151652. eCollection 2016. PMID 27011355